CLINICAL TRIAL: NCT05314777
Title: Comparison of the Efficacy of Extracorporeal Shock Wave Therapy (ESWT) at Different Pulse Numbers in Carpal Tunnel Syndrome
Brief Title: Efficacy of Extracorporeal Shock Wave Therapy in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Karaaslan, Ph.D. Pt., University of Beykent
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 02032022
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Extracorporeal Shockwave Therapy; Median Neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose ESWT application group (Experimental): Exercise Training Low dose ESWT application
  Interventions: Procedure: Low dose ESWT application; Procedure: Exercise Training
- High dose ESWT group (Experimental): Exercise Training High dose ESWT application
  Interventions: Procedure: High dose ESWT application; Procedure: Exercise Training
- Control group (Active Comparator): Exercise Training Sham ESWT
  Interventions: Procedure: Sham ESWT; Procedure: Exercise Training

INTERVENTIONS:
Procedure: Low dose ESWT application — Patients trained for low dose ESWT application.
  Arms: Low dose ESWT application group
Procedure: High dose ESWT application — Patients trained for high dose ESWT application.
  Arms: High dose ESWT group
Procedure: Sham ESWT — Patients trained for sham ESWT.
  Arms: Control group
Procedure: Exercise Training — Patients trained for exercise training.

SUMMARY:
The aim of the study is to examine the effects of ESWT applications at different pulse rates on pain, function, grip strength and median nerve conduction velocity in patients with Carpal Tunnel Syndrome. The patients will be randomly divided into 3 groups: the low dose ESWT group (28), the high dose ESWT group (28), and the control group (28). The first two groups will receive ESWT treatment at different doses, while the control group will be treated with sound only (1 time/week-3 weeks).

DETAILED DESCRIPTION:
The aim of the study is to examine the effects of ESWT applications at different pulse rates on pain, function, grip strength and median nerve conduction velocity in patients with Carpal Tunnel Syndrome. The sample of the study will consist of patients with carpal tunnel syndrome who were diagnosed in Gaziosmapaşa Training and Research Hospital between April 2022 and December 2022 and whose symptoms have persisted for at least 3 months. The patients will be randomly divided into 3 groups: the low dose ESWT group (28), the high dose ESWT group (28), and the control group (28). The first two groups will receive ESWT treatment at different doses, while the control group will be treated with sound only (1 time/week-3 weeks). The evaluation of the patients participating in the study will be made by the physician who is not aware of the groups. Evaluations will be made 3 times before the treatment, at the 1st month and at the 3rd month. In the evaluation, Boston Carpal Tunnel Syndrome Questionnaire to evaluate symptoms and functionality, visual analog scale (VAS) to evaluate pain, SF-36 to evaluate quality of life, hand dynamometer to evaluate grip strength and electrodiagnostic examination to evaluate median nerve conduction velocity will be performed. After the initial evaluations, the patients participating in the study will be randomly divided into 3 groups. Tendon shifting and nerve shifting exercises will be performed in all groups. ESWT will be applied to 2 groups at different beat numbers. One session of ESWT will be applied to both groups each week for 3 consecutive weeks. In addition to the exercises in the low dose ESWT group, 1000 beats at a pressure of 4 bar and a frequency of 5 Hz will be applied on the ESWT carpal tunnel. In addition to the exercises in the high-dose ESWT group, 2000 beats at a pressure of 4 bar and a frequency of 5 Hz will be applied on the ESWT carpal tunnel. In the control group, in addition to the exercises, sham ESWT will be applied. No energy will be used in Sham ESWT application, only sound will be given. Each group will be given a 15-minute cold-pack application after the ESWT application. The exercises will be taught to the patient before the first ESWT application and the exercises will be given to the patients in brochure form. These exercises will be given to the patient as home exercises. You will be asked to do these exercises at home in 2 sets of 5 repetitions 2 times a day. Tendon gliding exercises are performed with the fingers in 5 different positions as regular grip, hook grip, fist, desktop and normal fist. In the distal median nerve gliding exercise, firstly, in the neutral position of the wrist, the fingers and thumb are flexed, in the second position, all the fingers are in the neutral position, in the third position, when the thumb is in the neutral position, the wrist and other fingers are in extension, in the fourth position, the wrist, thumb and other fingers are in extension, In the fifth position, when the wrist and fingers are in the same position, the forearm is in supination, in the sixth position, in the fifth position, the thumb stretching is applied.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 18-65,

* Clinical symptoms persisting for at least 3 months
* Pain, tingling and paresthesia in the first 3 fingers together with the Phalen and Tinel test makes the patient positive,
* Patients who are positive are evaluated by a specialist in electrodiagnostic testing and the clinical stage of CTS is determined.
* Mild to moderate CTS is diagnosed if the sensory nerve action potential (SNAP) is >6 μV and the combined muscle action potential (CMAP) is >2.1 mV.
* Being diagnosed with mild and moderate CTS

Exclusion Criteria:

* The patient who received CTS operation or corticosteroid treatment,
* Presence of systemic diseases that will affect our treatment such as diabetes, rheumatoid arthritis, gout,
* It has been determined as atrophy in the thenar region of the hand (Xu,2020).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | First month- Third month
  The boston carpal tunnel syndrome questionnaire will be used to measure the severity of the disease and the level of functionality.

SECONDARY OUTCOMES:
Hand Grip Force | First month- Third month
  Hand grip strength will be measured with a Jamar dynamometer.
Nerve Conduction Velocity | First month- Third month
  The conduction velocity of the median nerve will be measured according to the American Academy of Neurology
Short Form- 36 | First month- Third month
  The quality of life of the patients will be evaluated with short form 36.
Visual analog scale | First month- Third month
  The pain intensity felt by the participants during rest and activity, respectively, will be evaluated by VAS

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Karaaslan, Ph.D., Principal Investigator — Beykent University; Fatih Ozyurt, Pt, Study Chair — Beykent University
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)